CLINICAL TRIAL: NCT07331922
Title: Landing Place: Impact of the Landing Place Mental Health App on Mental Health and Well-being
Brief Title: Mental Health App and Impact on Wellbeing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Christopher Shelton, PhD, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00024830
Record Dates: First submitted 2025-12-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Well-Being, Psychological
Keywords: Digital Mental Health; College Students; Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Group 1 will not use the app at all.
- App-intervention group (Experimental): Group 2 will use the mental health app almost every day for 4 weeks. The following activities must be completed in-app by participants in this arm:
  * Cognitive exercise (2 per week)
  * Mindfulness (2 per week)
  * Mood tracker (4 per week)
  * Chat feature (2 per week)
  * Articles (3 across the 4 weeks)
  * Journal (3 across the 4 weeks)
  * To-do (related to the goal, once a week)
  * Goals (1 goal at the beginning)
  Interventions: Behavioral: mental health app

INTERVENTIONS:
Behavioral: mental health app — The intervention will be the use of an AI-powered mental health app that includes activities based on evidence-based therapeutic techniques, mindfulness, goal setting, journaling, mood tracking, and educational material. The app is secure, easy-to-use, and customized for the needs of the college students.
  Arms: App-intervention group

SUMMARY:
The goal of this clinical trial is to learn if intervention with Landing Place mental health app can support wellness in college students. The main questions it aims to answer are:

Can the app increased well-being in college students? Will the app have increased use and usability by the college students? Researchers will compare two groups of participants to see if the app intervention will increase wellbeing and app usability rates.

Participants will randomly assigned into group 1 and 2. Group 1 will not use the app at all. Group 2 will use the app almost every day for 4 weeks.

DETAILED DESCRIPTION:
Mental health concerns across the United States have increased substantially, affecting individuals across age groups, geographic regions, and socioeconomic backgrounds. Emerging adults demonstrate the highest prevalence of mental health conditions among adult populations, while simultaneously exhibiting the lowest rates of treatment utilization. Barriers to treatment for this population include limited affordability, accessibility, availability, and acceptability of mental health services.

Digital mental health interventions have demonstrated effectiveness across a range of outcomes, including symptom reduction, self-management, and well-being enhancement. Smartphone-based applications, in particular, have been evaluated as tools to integrate mental health support through scalable and accessible technologies. Such applications may offer features including guided self-help activities, mindfulness practices, journaling, mood tracking, psychoeducational content, and location-based resources for mental health services.

Following the COVID-19 pandemic, mental health challenges among U.S. college students have intensified, with documented impacts on academic performance and overall functioning. These challenges are further exacerbated by stigma, financial constraints, and limited access to campus-based or community mental health services, particularly for students from historically marginalized backgrounds.

In response to these needs, Penn State Behrend's Virtual/Augmented Reality (VAR) Lab developed the Landing Place mental health app, a free digital intervention designed to support mental wellness among college students in the Erie region. The application was developed with an emphasis on usability, privacy, and accessibility, and is tailored to the developmental and contextual needs of young adults. Planned future iterations of the application aim to extend its use to additional populations, such as survivors of domestic violence.

The Landing Place app incorporates artificial intelligence, supported features and evidence-based therapeutic components, including mindfulness exercises, goal-setting activities, journaling, mood tracking, and educational content related to mental health and coping strategies. This clinical trial evaluates the effectiveness, usability, and acceptability of the application when used as a self-guided mental wellness intervention among college students.

The study examines multiple forms of data, including behavioral change measures, user engagement metrics, usability assessments, and participant feedback, to assess the app's utility in supporting well-being. It is hypothesized that participants who use the application will demonstrate increased well-being compared to a control group, along with higher engagement and acceptability of the app-based intervention modality.

ELIGIBILITY:
Inclusion Criteria:

* Penn State Behrend students
* Over the age of 18
* Must have an iPhone

Exclusion Criteria:

* People outside of Penn State
* Minors
* People currently in therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Well-being related to Attention and Cognitive Functioning | From enrollment to the end of intervention at 5 weeks
  Attention-related symptoms will be assessed using the DSM-5-TR Attention-Deficit/Hyperactivity Disorder and Sluggish Cognitive Tempo Measure, a self-report scale evaluating attentional functioning. Scores vary by subscale, with higher scores indicating greater symptom severity.
Well-being related to Health-related quality of life | From enrollment to the end of the intervention at 5 weeks
  Health-related quality of life will be measured using the Medical Outcomes Study Short Form-36 Health Survey (SF-36). The instrument generates domain scores ranging from 0 to 100, with higher scores indicating better perceived health and well-being.
Well-being related to Mental Health Symptom Severity | From enrollment to the end of the intervention at 5 weeks
  Mental health symptom severity will be assessed using the Depression Anxiety Stress Scales - 21 Items (DASS-21), a self-report instrument measuring symptoms of depression, anxiety, and stress. Scores range from 0 to 63, with higher scores indicating greater symptom severity.
Well-being related to Functional Impairment | From enrollment to the end of the intervention at 5 weeks
  Functional impairment will be evaluated using the Brief Functional Impairment Scale - Long Form (BFIS-LF), which assesses impairment across daily functioning domains. Scores range from 0 to 100, with higher scores indicating greater functional impairment.

SECONDARY OUTCOMES:
Usability | From enrollment to the end of treatment at 5 weeks
  App usability will be assessed using the mHealth App Usability Questionnaire - Standalone Patient App Version (MAUQ-SPA), a self-report instrument designed to evaluate the usability of standalone mHealth applications. Items are rated on a 7-point Likert scale, and total scores range from 1 to 7, with higher scores indicating better perceived usability.
Usage | From enrollment to the end of the intervention at 5 weeks
  Patterns of mobile health application use will be assessed using the mHealth Usage Questionnaire, a self-report measure evaluating frequency and duration of app use. Scores are reported in units on a scale, with higher scores indicating greater application use.
Engagement | From enrollment to the end of the intervention at 5 weeks
  Engagement with mobile health technology will be measured using the mHealth Technology Use Questionnaire, which assesses overall use and engagement with mHealth technologies. Scores are reported in units on a scale, with higher scores indicating greater technology engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- PennState the Beherend College/VAR Lab, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: IPD will be shared with qualified researchers upon submission of a scientifically sound research proposal. Requests must include a description of the research objectives and planned analyses and must be consistent with the original informed consent and applicable ethical approvals. Access to the data will be granted following review of the proposal for scientific and methodological appropriateness. Approved requestors will be required to sign a data sharing agreement that outlines the conditions for data use, data security, confidentiality, and publication. De-identified data will be made available in a secure manner and will be used solely for the purposes approved.

REFERENCES:
- [Background] Andersson, G., & Titov, N. (2014). Advantages and limitations of Internet-based interventions for common mental disorders. World Psychiatry; Official Journal of the World Psychiatric Association (WPA), 13(1), 4-11. doi:10.1002/wps.20083 PMID:24497236 Barak, A., Hen, L., Boniel-Nissim, M., & Shapira, N. (2008). A comprehensive review and a meta-analysis of the effectiveness of internet-based psychotherapeutic interventions. Journal of Technology in Human Services, 26(2-4), 109-160. doi:10.1080/15228830802094429 Boggs, J. M., Beck, A., Felder, J. N., Dimidjian, S., Metcalf, C. A., & Segal, Z. V. (2014). Web-Based Intervention in Mindfulness Meditation for Reducing Residual Depressive Symptoms and Relapse Prophylaxis: A Qualitative Study. Journal of Medical Internet Research, 16(3), e87. doi:10.2196/jmir.3129 PMID:24662625 Hedman, E., El Alaoui, S., Lindefors, N., Andersson, E., Rück, C., Ghaderi, A., Kaldo, V., Lekander, M., Andersson, G., & Ljótsson, B. (2014). Clinical effectiveness and cost-effectiveness of Internet- vs. group-based cognitive behavior therapy for social anxiety disorder: 4-year follow-up of a randomized trial. Behaviour Research and Therapy, 59, 20-29. doi:10.1016/j.brat.2014.05.010 PMID:24949908 Luxton, D. D., McCann, R. A., Bush, N. E., Mishkind, M. C., & Reger, G. M. (2011). mHealth for mental health: Integrating smartphone technology in behavioral healthcare. Professional Psychology, Research and Practice, 42(6), 505-512. doi:10.1037/a0024485 Proudfoot, J. G. (2004). Computer-based treatment for anxiety and depression: Is it feasible? Is it effective? Neuroscience and Biobehavioral Reviews, 28(3), 353-363. doi:10.1016/j.neubiorev.2004.03.008 PMID:15225977 Substance Abuse and Mental Health Services Administration. (2017). Key substance use and mental health indicators in the United States: Results from the 2016 National Survey on Drug Use and Health (HHS Publication No. SMA 17-5044, NSDUH Series H-52). Rockville, MD: Center for Behavioral